CLINICAL TRIAL: NCT05197270
Title: A Phase 1/2 Dose-Escalation and Randomized, Controlled, Masked Expansion Trial of Intravitreal 4D-150 Gene Therapy in Adults With Neovascular (Wet) Age-Related Macular Degeneration
Brief Title: 4D-150 in Patients With Neovascular (Wet) Age-Related Macular Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 4D-150-C001
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neovascular (Wet) Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; Exudative AMD; Exudative age-related macular degeneration; Neovascular AMD; Neovascular age-related macular degeneration; Wet age-related macular degeneration; Wet macular degeneration; Wet AMD; wAMD; Retinal gene therapy; Intravitreal gene therapy; Genetic Medicine; Ocular Gene Therapy
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration

STUDY DESIGN:
Intervention Model Description: In Dose Escalation, the safety and tolerability of multiple dose levels of 4D-150 will be examined following an open-label, 3+3 dose escalation design (n=3-5 per dose level). In Dose Expansion, subjects (n=50) will be randomized to receive one of 2 dose levels of 4D-150 (n=20 for each dose level) based on results from Dose Escalation, or aflibercept (n=10). In Steroid Optimization (n=up to 96) and Population Extension (n=up to 45) Cohorts, subjects will be assigned sequentially to receive 4D-150 at doses cleared by the DSMC.
  Contralateral sub-study: Up to 20 subjects from the 4D-150-C001 trial who have previously received 4D-150 in study eye-1 will be enrolled and administered a single open-label IVT injection of 4D-150 in the contralateral eye.
  Vector Shedding sub-study: Approximately 15 subjects will receive an open-label IVT injection of 4D-150 to evaluate vector shedding.
Who Masked: Outcomes Assessor
Masking Description: Dose Escalation will be open-label. During Dose Expansion, outcome assessors will be masked to treatment assignment. Other site personnel (including investigator) and subjects will be unmasked to treatment assignment but will be masked to 4D-150 dose level. The Sponsor and its representatives and the site dose preparer/pharmacist will be unmasked to treatment assignment. Steroid Optimization and Population Extension will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- 4D-150 Dose Escalation up to 4 dose levels (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Dose Expansion Dose 1 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Dose Expansion Dose 2 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Dose Expansion Control (Active Comparator): Aflibercept at a fixed regimen will be administered.
  Interventions: Biological: Aflibercept IVT
- 4D-150 Steroid Optimization (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Population Extension Dose 1 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Population Extension Dose 2 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Population Extension Dose 3 (Experimental): 4D-150 will be administered at the assigned dose
  Interventions: Biological: 4D-150 IVT
- 4D-150 Contralateral Eye Dose (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Vector Shedding Dose (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT

INTERVENTIONS:
Biological: 4D-150 IVT — 4D-150: AAV-based gene therapy comprised of miRNA targeting VEGF-C and codon-optimized sequence encoding aflibercept
  Arms: 4D-150 Contralateral Eye Dose; 4D-150 Dose Escalation up to 4 dose levels; 4D-150 Dose Expansion Dose 1; 4D-150 Dose Expansion Dose 2; 4D-150 Population Extension Dose 1; 4D-150 Population Extension Dose 2; 4D-150 Population Extension Dose 3; 4D-150 Steroid Optimization; 4D-150 Vector Shedding Dose
Biological: Aflibercept IVT — Commercially available Active Comparator Other Name: Eylea
  Arms: 4D-150 Dose Expansion Control

SUMMARY:
Phase 1/2 dose-escalation and randomized, controlled, masked expansion trial in adults with wet AMD undergoing active anti-VEGF treatment.

Substudies will evaluate the safety and tolerability of 4D-150 contralateral eye dosing and characterize vector shedding.

DETAILED DESCRIPTION:
This Phase 1/2 trial is a prospective, multicenter, Phase 1/2 dose-escalation and randomized, controlled, masked expansion trial in adults with wet AMD undergoing active anti-VEGF treatment who have demonstrated a clinical response consistent with anti-VEGF activity. The trial consists of Dose Escalation, Dose Expansion, Steroid Optimization, and[DD1.1][JA1.2] Population Extension Cohorts.

After receiving one time administration of 4D-150 by intravitreal injection (IVT), subjects will undergo assessments at monthly intervals for 24 months to assess safety and efficacy outcomes. Only subjects that received 4D-150 will then enter a long-term follow-up (LTFU) period to assess long-term safety of 4D-150 gene therapy and duration of clinical activity through year 5 (60 months).

Eligible subjects who received 4D-150 in the study eye may participate in a sub-study to evaluate one-time IVT administration of 4D-150 to the contralateral ("fellow") eye.

Additional subjects will be enrolled in a separate sub-study to characterize the vector shedding profile of one-time administration of IVT 4D-150.

In both sub-studies, subjects will undergo regular assessments to assess safety and tolerability through Week 52 and then will enter long-term follow-up for safety evaluation through year 5 (60 months).

ELIGIBILITY:
* 50 years of age

Individuals eligible to participate in the trial must meet the following inclusion criteria:

1. ≥50 years of age
2. Diagnosed with CNV secondary to AMD (confirmed by reading center)
3. BCVA ≥34 ETDRS letters (~20/200) in the contralateral eye, and BCVA in the study eye:
4. Central subfield thickness (CST) and/or presence of subretinal or intraretinal fluid requiring continued anti-VEGF therapy in the study eye, as assessed by SD-OCT; and confirmed by a reading center):
5. Study eye amenable to IVT injection
6. Ability to perform tests of visual and retinal function and structure, and ability to comply with other protocol-specified procedures
7. Currently receiving anti-VEGF treatment (e.g. ranibizumab, aflibercept, faricimab or bevacizumab) in the study eye AND has demonstrated a clinical response consistent with anti-VEGF activity within 12 months prior to screening:

   Note: Day -7 aflibercept will be administered ≥ 4 weeks from last IVT anti-VEGF
8. Subjects receiving 4D-150 agree to use a barrier method (e.g. condom) during intercourse for 6 months after administration of 4D-150 to prevent fluid transmission; sexually active males should not father a child or donate sperm during this period
9. Medical records available to document history of anti-VEGF therapy (dates, drugs, and dosage) for a minimum of 12 months prior to Screening
10. Provide written informed consent.

Contralateral Eye Sub-study-Specific Criteria:

1. Received 4D-150 in study eye-1 at least 6 months prior to Contralateral Substudy Screening Visit NOTE: Subjects who received 4D-150 in study eye-1 as part of the Shedding Substudy are also eligible to participate in the Contralateral Eye Substudy only after biological samples from all matrices were at or below the limit of quantitation for vector genomes in at least 3 consecutive measurements AND at least 6 months has passed since 4D-150 administration to study eye-1.
2. Macular neovascularization (MNV) secondary to AMD in study eye-2 as assessed on historical images at any time by SD-OCT (required) and FA when available or fundus photography when available or at screening based on SD-OCT, FA and fundus photography (confirmed by the reading center)
3. History of at least 1 anti-VEGF injection in study eye-2 within 6 months prior to Screening (last anti-VEGF injection must be at least 28 days prior to Screening) AND has demonstrated a clinical response consistent with anti-VEGF activity by historical OCT at any time point prior to screening with confirmed response by the reading center (Screening OCT can be confirmatory)
4. BCVA between 25 and 83 ETDRS letters, inclusive (20/320 20/25 Snellen) in study eye-2
5. Study eye-2 amenable to IVT injection
6. BCVA ≥34 ETDRS letters (~20/200) in the previously treated study eye-1
7. Ability to comply with protocol-specified procedures and visits, in the Investigator's judgment
8. Agree to use a barrier method (e.g. condom) during intercourse for 6 months after administration of 4D-150 to study eye-2 to prevent fluid transmission; sexually active males should not father a child or donate sperm during this period
9. Provide written informed consent.

Shedding Substudy-specific Inclusion Criteria:

1. ≥50 years of age
2. Diagnosed with MNV secondary to AMD as assessed on historical images at any time by spectral domain optical coherence tomography (SD-OCT) (required) and fluorescein angiography when available or fundus photography when available or at screening based on SD-OCT, FA and fundus photography (confirmed by Reading Center)
3. Best corrected visual acuity (BCVA) between 10 and 83 ETDRS letters, inclusive (~20/640 and 20/25, respectively) in the study eye at Screening
4. BCVA ≥34 ETDRS letters (~20/200) in the contralateral eye
5. Currently receiving anti-VEGF treatment (e.g. ranibizumab, aflibercept, faricimab or bevacizumab) in the study eye; minimum of 1 injection within the last 6 months (last anti-VEGF injection must be at least 28 days prior to screening) AND has demonstrated a clinical response consistent with anti-VEGF activity by historical OCT at any time prior to screening with confirmed response by the reading center (Screening OCT can be confirmatory)
6. Study eye amenable to IVT injection
7. Ability to perform tests of visual and retinal function and structure, and ability to comply with other protocol-specified procedures, in the Investigator's judgment
8. Agree to use a barrier method (e.g. condom) during intercourse for 6 months after administration of 4D-150 to prevent fluid transmission; sexually active males should not father a child or donate sperm during this period
9. Provide written informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs), including clinically significant changes in safety parameters | 52 weeks

SECONDARY OUTCOMES:
Time to receiving the first supplemental aflibercept injection | 52 weeks
Percentage of subjects requiring supplemental aflibercept injections over 52 weeks | 52 weeks
Number of supplemental aflibercept injections over 52 weeks | 52 weeks
Change from baseline in BCVA over time (up to 52 weeks) as assessed using the ETDRS Visual Acuity Chart | 52 weeks
Change from baseline in central subfield thickness (CST) over time (up to 52 weeks) measured by spectral domain optical coherence tomography (SD-OCT) | 52 weeks
Percent Change in Annualized Mean Number of anti-VEGF IVT injections before and after the 4D-150 injection | Before and after the 4D-150 injection (or Day 1 for the aflibercept only arm)
  Percent change in annualized mean number of anti-VEGF IVT injections before and after the 4D-150 injection (or Day 1 for the aflibercept only arm)

CONTACTS AND LOCATIONS:
Overall Officials: Demi Dang, MD, Study Director — 4D Molecular Therapeutics
Locations (25):
- United States (24):
  - Barnet Delaney Perkins Eye Center, Phoenix, Arizona
  - California Retina Consultants, Oxnard, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Colorado Retina Associates, Lakewood, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Vitreous Consultants, LLP DBA Retina Group of Florida, Fort Lauderdale, Florida
  - Vitreo Retinal Associates, Gainesville, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retinal Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Retina Partners Midwest, Carmel, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston & Boston Eye Surgery and Laser Center, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Verum Research, LLC, Eugene, Oregon
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - Tennessee Retina, Nashville, Tennessee
  - Austin Clinical Research, Austin, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Pacific Northwest Retina LLC, Bellevue, Washington
- Emanuelli Research and Development Center, LLC, Arecibo, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No